CLINICAL TRIAL: NCT03307096
Title: Evaluation of Two Different Treatments for Lower Pore Renal Stone: Microperc Vs FURS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The project has come to an end due to a lack of necessary funding support.
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Renmin Hospital of Wuhan University (Other); Affiliated Hospital of Hebei University (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); West China Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); People's Hospital of Anshun City of Guizhou Province (Other); Zhejiang Provincial People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Li Fang, Urologist, Ningbo No. 1 Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NBDYYY2017003
Record Dates: First submitted 2017-09-30; First posted 2017-10-11 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Surgery--Complications; Renal Calculus; Nephrolithiasis; Urolithiasis
Keywords: FURS; microperc; renal calculus; Randomized Controlled Trial; Retrograde Intrarenal Surgery
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Intervention Model Description: A total of 200 patients, aging between 18 and 60 years are enrolled into the study, patients will be prospectively randomized into group A and group B with a 1:1 ratio. Group A will receive the microperc surgery and group B will undergo FURS.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microperc surgery (Experimental): Patient is turned into prone position and the desired calyx is punctured by 4.8F microperc under fluoroscopic or sonographic guidance. No tract dilation is needed. A 200um holmium laser fiber will be used to break stone into less than 2mm. Pull out microperc without drainage tube left.
  Interventions: Procedure: Microperc surgery
- FURS (Active Comparator): Patient is placed in the lithotomy position, pull out the pre-inserted double J, and place guidewire into the renal pelvis. A 12/14 Fr ureteral access sheath (UAS) is advanced into the proximal ureter over the guidewire, and flexible ureteroscope is passed through the UAS. The stones are fragmented smeller than 2mm using a 200um holmium laser fiber. Fragments are removed using a stone basket for stone analysis if necessary, a double J stent is placed at the conclusion of the procedure and removed post-operative 4 weeks.
  Interventions: Procedure: FURS

INTERVENTIONS:
Procedure: Microperc surgery — Parents are treated by Microperc Percutaneous Nephrolithotomy
  Arms: Microperc surgery
Procedure: FURS — Parents are treated by FURS
  Arms: FURS

SUMMARY:
This is a prospect, randomized control trial to evaluate merits between microperc and FURS for lower pole renal stone

DETAILED DESCRIPTION:
To evaluate the merits of Microperc and RIRS for the treatment for lower pole renal stone between 10-20 mm. Investigators will do a multi-centers randomized controlled trial(RCT). A total of 200 (three hundred) patients, aging between 18 and 60 years are being planned to be enrolled into the study; By simple random sampling technique, patients will be prospectively randomized into group A and group B with a 1:1 ratio. Group A will receive the microperc surgery and group B will undergo FURS.

All the patients will be diagnosed definitely before operations with non-contrast CT+IVP or CTU, lower pole Infundibular length, Infundibular width and Lower pole infundibulopelvic angle were recorded. A double J stent will be inserted in two the relevant ureter two weeks before surgery to guarantee the successful of operations. Patience will receive either microperic or FURS respectively, The operation time , hemoglobin change, renal function, post-operation pain, complications and hospital stay will be recorded. Patience will have follow-up visits at one month and three months, CT and KUB will be taken to evaluate the clearance of renal stone.

Surgical technique Microperc surgery: After the satisfaction of anesthesia, Patient is turned into prone position and the desired calyx is punctured by 4.8F microperc under fluoroscopic or sonographic guidance. No tract dilation is needed. A 200um holmium laser fiber will be used to break stone into less than 2mm. Pull out microperc without drainage tube left; RIRS: After the satisfaction of anesthesia, the patient is placed in the lithotomy position, pull out the pre-inserted double J stent, and place guidewire into the renal pelvis. A 12/14 Fr ureteral access sheath (UAS) is advanced into the proximal ureter over the guidewire, and flexible ureteroscope is passed through the UAS. The stones are fragmented smeller than 2mm using a 200um holmium laser fiber. Fragments are removed using a stone basket for stone analysis if necessary, a double J stent is placed at the conclusion of the procedure and removed post-operative 2 weeks.

Data collection Data for the 2 groups-demographic characteristics, hemoglobin(HB) decrease, white blood cell(WBC) increase, postoperative pain, duration of postoperative hospital stay, complications (modified Clavien system), stone clearance (SFR) and the need for auxiliary treatment are compared.

Mean study endpoint: Final SFR (3 months after procedure) Secondary endpoint: Complications, duration of postoperative hospital stay. re-microperc, ureteroscopy and SWL are considered as auxiliary treatments.

The stone size is defined as the maximum diameter as determined by CT scans. Degree of hydronephrosis are assigned as follow: none (no calyx or pelvic dilation), mild (pelvic dilatation alone), moderate (mild calyx dilation), or severe (severe calyx dilation or calyx dilation accompanied by renal parenchyma atrophy).

Definition of operation time:

For microperc: recorded from the time of the first percutaneous renal puncture to pulling out the microperc.

For RIRS: recorded from insertion of an endoscope into the urethra to the completion of stent placement.

Hospital stay are rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.

Postoperative pain (visual analogue scale(VAS), use of analgesics) will be recorded.

The rate of hemoglobin decrease is assessed by comparing the preoperative Hb level with 24-hour postoperative Hb level.

Non-contrast CT and KUB is obtained for all patients at 3 month after the operation to evaluate the final SFR, allowing time for the spontaneous passage of stone fragments.

Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≤4mm, asymptomatic, non-obstructive and non-infectious stone particles.

Complications of all patients are recorded according to modified Clavien classification system.

ELIGIBILITY:
Inclusion Criteria:

1. 10-20mm lower pole renal stone measured by KUB or CT;
2. Age between 18-60 years, no gender limitation;
3. Participators can understand the research and sign the consent form without mental illness nor language disorder;
4. Low pole renal stone left after lithotripsy;
5. Lower pole infundibulopelvic angle which measured by IVP or CTU will less than 30 degree;
6. Asymptomatic patients with positive urine white blood cells and negative preoperative urine culture should be treated with antibiotics for 3days before operation;
7. Patients with symptoms of urinary infections, positive urine withe blood cells and positive preoperative urine culture should be treated with suitable antibiotics based on the culture sensitivity result for at least 7days before operation.

Exclusion Criteria:

1. Transplant kidney stone;
2. Renal malformations, such as UPJO, medullary sponge kidney, polycystic kidney, horseshoe kidney, etc.;
3. Combine other part of urinary stones need to be handle at the same procedure, for example ureteral stone, renal pelvic stone, middle or upper pole renal stone;
4. Hematological Disease or Coagulation disorders;
5. Withdraw anticoagulant medicine less than two weeks;
6. Fever or urinary infections without treatment according to the inclusion criteria;
7. Sevier renal dysfunction(endogenous creatinine clearance rate≤50ml/min)
8. Middle or severe hydronephrosis(dilatation of the renal pelvis ≥20mm by ultrasound);
9. Women in menstrual period or pregnancy;
10. Patients have severe disease, such as heart disease, lung dysfunction, and multiple organ failure that cannot tolerate anesthesia or operation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-17 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
SFR | 3 month
  Stone free Rate

SECONDARY OUTCOMES:
Complications | 3 month
  Complications after surgery
Duration of postoperative hospital stay | 7 days
  Duration of postoperative hospital stay
Postoperative pain | 3 month
  Postoperative pain,visual analogue scale(VAS)
The rate of hemoglobin decrease | 7 days
  The rate of hemoglobin decrease
Operation time | 12 hours
  Operation time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yue Cheng, Dr., Principal Investigator — Ningbo No. 1 Hospital
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sener NC, Imamoglu MA, Bas O, Ozturk U, Goktug HN, Tuygun C, Bakirtas H. Prospective randomized trial comparing shock wave lithotripsy and flexible ureterorenoscopy for lower pole stones smaller than 1 cm. Urolithiasis. 2014 Apr;42(2):127-31. doi: 10.1007/s00240-013-0618-z. Epub 2013 Nov 13. PMID 24220692
- [Background] Ozgur Tan M, Irkilata L, Sen I, Onaran M, Kupeli B, Karaoglan U, Bozkirli I. The impact of radiological anatomy in clearance of lower caliceal stones after shock wave lithotripsy. Urol Res. 2007 Jun;35(3):143-7. doi: 10.1007/s00240-007-0093-5. Epub 2007 Apr 20. PMID 17447057
- [Background] Juan YS, Chuang SM, Wu WJ, Shen JT, Wang CJ, Huang CH. Impact of lower pole anatomy on stone clearance after shock wave lithotripsy. Kaohsiung J Med Sci. 2005 Aug;21(8):358-64. doi: 10.1016/S1607-551X(09)70134-2. PMID 16158878
- [Background] Turk C. [Urolithiasis guidelines: retrospective view and perspectives]. Urologe A. 2016 Oct;55(10):1317-1320. doi: 10.1007/s00120-016-0230-2. German. PMID 27604704
- [Background] Molina WR, Kim FJ, Spendlove J, Pompeo AS, Sillau S, Sehrt DE. The S.T.O.N.E. Score: a new assessment tool to predict stone free rates in ureteroscopy from pre-operative radiological features. Int Braz J Urol. 2014 Jan-Feb;40(1):23-9. doi: 10.1590/S1677-5538.IBJU.2014.01.04. PMID 24642147
- [Background] Elbahnasy AM, Clayman RV, Shalhav AL, Hoenig DM, Chandhoke P, Lingeman JE, Denstedt JD, Kahn R, Assimos DG, Nakada SY. Lower-pole caliceal stone clearance after shockwave lithotripsy, percutaneous nephrolithotomy, and flexible ureteroscopy: impact of radiographic spatial anatomy. J Endourol. 1998 Apr;12(2):113-9. doi: 10.1089/end.1998.12.113. PMID 9607435
- [Result] Resorlu B, Unsal A, Gulec H, Oztuna D. A new scoring system for predicting stone-free rate after retrograde intrarenal surgery: the "resorlu-unsal stone score". Urology. 2012 Sep;80(3):512-8. doi: 10.1016/j.urology.2012.02.072. Epub 2012 Jul 26. PMID 22840867
- [Result] Kilicarslan H, Kaynak Y, Kordan Y, Kaygisiz O, Coskun B, Gunseren KO, Kanat FM. Unfavorable anatomical factors influencing the success of retrograde intrarenal surgery for lower pole renal calculi. Urol J. 2015 Apr 29;12(2):2065-8. PMID 25923149
- [Result] Resorlu B, Oguz U, Resorlu EB, Oztuna D, Unsal A. The impact of pelvicaliceal anatomy on the success of retrograde intrarenal surgery in patients with lower pole renal stones. Urology. 2012 Jan;79(1):61-6. doi: 10.1016/j.urology.2011.06.031. PMID 21855968
- [Result] Inoue T, Murota T, Okada S, Hamamoto S, Muguruma K, Kinoshita H, Matsuda T; SMART Study Group. Influence of Pelvicaliceal Anatomy on Stone Clearance After Flexible Ureteroscopy and Holmium Laser Lithotripsy for Large Renal Stones. J Endourol. 2015 Sep;29(9):998-1005. doi: 10.1089/end.2015.0071. Epub 2015 May 15. PMID 25879676
- [Result] Sabnis RB, Ganesamoni R, Doshi A, Ganpule AP, Jagtap J, Desai MR. Micropercutaneous nephrolithotomy (microperc) vs retrograde intrarenal surgery for the management of small renal calculi: a randomized controlled trial. BJU Int. 2013 Aug;112(3):355-61. doi: 10.1111/bju.12164. PMID 23826843
- [Result] Karatag T, Tepeler A, Silay MS, Bodakci MN, Buldu I, Daggulli M, Hatipoglu NK, Istanbulluoglu MO, Armagan A. A Comparison of 2 Percutaneous Nephrolithotomy Techniques for the Treatment of Pediatric Kidney Stones of Sizes 10-20 mm: Microperc vs Miniperc. Urology. 2015 May;85(5):1015-1018. doi: 10.1016/j.urology.2015.02.010. PMID 25917724
- [Derived] Soderberg L, Ergun O, Ding M, Parker R, Borofsky MS, Pais V, Dahm P. Percutaneous nephrolithotomy versus retrograde intrarenal surgery for treatment of renal stones in adults. Cochrane Database Syst Rev. 2023 Nov 13;11(11):CD013445. doi: 10.1002/14651858.CD013445.pub2. PMID 37955353